CLINICAL TRIAL: NCT04392427
Title: Effect of a Combination of Nitazoxanide, Ribavirin and Ivermectin Plus Zinc Supplement on the Clearance of COVID-19: a Pilot Sequential Clinical Trial
Brief Title: New Antiviral Drugs for Treatment of COVID-19
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Hatem Elalfy, Professor of Tropical Medicine and Hepatogastroenterology, Mansoura University
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: 20.05.69
Record Dates: First submitted 2020-05-12; First posted 2020-05-18 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2020-09

CONDITIONS: COVID; Drug Effect
Keywords: COVID-19;; clinical trial; corona virus
MeSH Terms: conditions — COVID-19 | interventions — Ribavirin; Ivermectin

STUDY DESIGN:
Intervention Model Description: a sequential clinical trial in this design sample size is not fixed in advance. Instead data will be evaluated as they are collected, and further sampling is will be stopped in accordance with a pre-defined stopping rule as soon as significant results are observed. After "n" (10 subjects in each group) subjects in each group are available an interim analysis will be conducted. A statistical test will be performed to compare the two groups and if the null hypothesis is rejected the trial is terminated; otherwise, the trial continues, another n subjects per group will be recruited, and the statistical test is performed again, including all subjects. If the null is rejected, the trial is terminated, and otherwise it continues with periodic evaluations until a maximum number of interim analyses have been performed, at which point the last statistical test is conducted and the trial is discontinued
Who Masked: Outcomes Assessor
Masking Description: This search will focus on patients with COVID 19 infection this study is a prospective cohort study based on the analysis of response in comparative panel between two arm Nitazoxanide, Ribavirin and Ivermectin plus Zinc arm and other arm without any intervention as regards the safety and efficacy and cost effective result. Two years duration of the project would be enough to cover the stages of the work as shown below in the time plan. Initial stage of collecting materials and patients' clinical data, each patient will undergoes strict follow up period to reveal the clinical, laboratory and radiological response. The procedures are to be approved by the institutional ethical committee.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- INTERVENTION (Active Comparator): *Intervention:
  A) Treatment group: will receive a combination of Nitazoxanide, Ribavirin and Ivermectin for a duration of seven days :
  Interventions: Drug: Treatment group: will receive a combination of Nitazoxanide, Ribavirin and Ivermectin for a duration of seven days :
- CONTROL (No Intervention): B) Control group: will not receive nothing
  * Data collection will include: sociodemographic data, clinical history, results of follow up (daily or according to clinical situation )
  * Follow-up: to record any side effects of drugs, swab will be taken for PCR

INTERVENTIONS:
Drug: Treatment group: will receive a combination of Nitazoxanide, Ribavirin and Ivermectin for a duration of seven days : — Target population: any subject with COVID-19 PCR positive pharyngeal swab and referred to the above-mentioned quarantine without any comorbidities and no sensitivity or contraindication to the three drugs.
  * Sample size: will depends on sequential analysis until a significant effect will be detected with a maximum of 100 subjects in each arm.
  * Randomization: subjects will be allocated to either arm by block randomization method with sealed opaque envelops. Each block will include 10 subjects (to be allocated randomly as 5 in each group)
  * Intervention:
  A) Treatment group: will receive a combination of Nitazoxanide, Ribavirin and Ivermectin for a duration of seven days
  Other Names: Nanozoxide, ivermectin and ribavirin 200 mg or 400 mg
  Arms: INTERVENTION

SUMMARY:
Background: In December 2019, SARS-CoV-2 was isolated on Vero E6 and Huh7 cell lines after an outbreak of pneumonia of unknown origin in Wuhan, Hubei Province, China. Since the basis for pathogenesis of this virus and its proliferation is unclear, there is still no definitive treatment or vaccine against it. Thus, medications used against SARS-CoV-2 are mainly based on their effectiveness on in vitro studies, virtual screenings and records of their effects on earlier strains of coronavirus, SARS and MERS. Therefore, the immediate introduction of potential COVID-19 treatments can be essential and salvaging. Aim: to compare the rate and time of viral clearance in subjects receiving the combination of Nitazoxanide, Ribavirin and Ivermectin vs. those control group (without any intervention). Methods: a sequential clinical trial in this design sample size is not fixed in advance. Instead data will be evaluated as they are collected, and further sampling is will be stopped in accordance with a pre-defined stopping rule as soon as significant results are observed. After "n" (10 subjects in each group) subjects in each group are available an interim analysis will be conducted. A statistical test will be performed to compare the two groups and if the null hypothesis is rejected the trial is terminated; otherwise, the trial continues, another n subjects per group will be recruited, and the statistical test is performed again, including all subjects. If the null is rejected, the trial is terminated, and otherwise it continues with periodic evaluations until a maximum number of interim analyses have been performed, at which point the last statistical test is conducted and the trial is discontinued [25]. Outcome: The combination of Nitazoxanide, Ribavirin, Ivermectin and Zinc could be effective in clearance of COVID 19.

KEY WOARD: COVID-19; clinical trial; corona virus

DETAILED DESCRIPTION:
* Research Design and Methodologies:

This search will focus on patients with COVID 19 infection this study is a prospective cohort study based on the analysis of response in comparative panel between two arm Nitazoxanide, Ribavirin and Ivermectin plus Zinc arm and other arm without any intervention as regards the safety and efficacy and cost effective result. Two years duration of the project would be enough to cover the stages of the work as shown below in the time plan. Initial stage of collecting materials and patients' clinical data, each patient will undergoes strict follow up period to reveal the clinical, laboratory and radiological response. The procedures are to be approved by the institutional ethical committee.

Study Design:

After obtaining informed consent from the subjects and IRB approval from Mansoura Faculty of Medicine.

Technical Design:

The proposed study will be hospital- based cross- sectional study.

Data collection tools and techniques:

1-Clinical work package: The aim of the Tropical Department in Mansoura University within WP1 is to implement surveillance, diagnostic and monitoring models for the disease management of patients with COVID 19 infection according to the current scientific evidence. They will evaluate the clinical usefulness of the application of therapeutic clinical trial, to improve the disease outcomes and reduce the costs of the disease burdens.

In brief, the approach will consist of the following steps:

1. Diagnosis of patient with COVID 19 infection by swab and PCR testing
2. Tailored therapeutic strategy in patients with COVID 19 infection undergoing treatment by nitazoxanide, Ribavirin and Ivermectin plus Zinc (this done in collaboration with biochemical department and Clinical Pathology department in Mansoura University).
3. Patients with the other group will not undergoes any intervention.
4. Specific laboratory analysis for COVID 19 RNA by Polymerase Chain Reaction in nasopharyngeal and oropharyngeal swabs will be don't to both groups.
5. Monitoring the treatment response in the follow up periods.

Description of work and role of participants:

Rationale of study: COVID-19 is an emerging infection with relatively high transmission rate from healthy carriers to their contacts. There is no known drug that eliminate the virus from the nasopharynx.

Study objectives: to compare the rate and time of viral clearance in subjects receiving the combination of Nitazoxanide, Ribavirin and Ivermectin vs. those control group (without any intervention) Study hypothesis: The combination of Nitazoxanide, Ribavirin, Ivermectin plus zinc supplement have higher rate of viral clearance at earlier time than the control group

Population and methods:

* Study locality: subject with proven COVID-infection admitted to quarantine centers of Mansoura University Hospitals
* Study design: a sequential clinical trial in this design sample size is not fixed in advance. Instead data will be evaluated as they are collected, and further sampling is will be stopped in accordance with a pre-defined stopping rule as soon as significant results are observed. After "n" (10 subjects in each group) subjects in each group are available an interim analysis will be conducted. A statistical test will be performed to compare the two groups and if the null hypothesis is rejected the trial is terminated; otherwise, the trial continues, another n subjects per group will be recruited, and the statistical test is performed again, including all subjects. If the null is rejected, the trial is terminated, and otherwise it continues with periodic evaluations until a maximum number of interim analyses have been performed, at which point the last statistical test is conducted and the trial is discontinued [25].
* Target population: any subject with COVID-19 PCR positive pharyngeal swab and referred to the above-mentioned quarantine without any comorbidities and no sensitivity or contraindication to the three drugs.
* Sample size: will depends on sequential analysis until a significant effect will be detected with a maximum of 100 subjects in each arm.
* Randomization: subjects will be allocated to either arm by block randomization method with sealed opaque envelops. Each block will include 10 subjects (to be allocated randomly as 5 in each group)
* Intervention:

A) Treatment group: will receive a combination of Nitazoxanide, Ribavirin and Ivermectin B) Control group: will not receive nothing

* Data collection will include: sociodemographic data, clinical history, results of follow up (daily or according to clinical situation )
* Follow-up: to record any side effects of drugs, swab will be taken for PCR

  2-Laboratory and investigational work package:

The patients are subjected to following laboratory workup:

Task 2-1: basic laboratory serum analysis for the following parameters: transaminases (AST, ALT), albumin, bilirubin, prothrombin time, complete blood picture, renal assessment (creatinine or clearance if needed), CRP, Oxygen saturation

Task 2-2: specific laboratory analysis ( if available case by case ):

Serum samples from each patient are collected for analysis at different time for detection of ferritin, triglycerides, LDH,

3-Invetigational radiology work package:

This package includes chest x ray and /or high resolution CT

ELIGIBILITY:
Inclusion Criteria:

* any subject with COVID-19 PCR positive pharyngeal swab and referred to the above-mentioned quarantine without any comorbidities and no sensitivity or contraindication to the three drugs.

Exclusion Criteria:

* PATIENTS WITH COMORBIDITY :ISCHEMIC HEART DISEASES,OR KNOWN HYPERSENSITIVITY TO THE DRUGS

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-10 (Estimated); Primary Completion 2022-05 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
negative test result for COVID-19 | 2 YEARS
  PCR FOR COVID-19 will be done on serial visits till turn to negative, first after 5 day then serial every 48 hours till become negative for two consecutive samples.

CONTACTS AND LOCATIONS:
Overall Officials: HATEM ELALFY, MD, Principal Investigator — PROFESSOR OF ENDEMIC MEDICINE DEPARTMENT; HATEM ELALFY, MD, Principal Investigator — Mansoura University
Locations (1):
- Mansoura University, Al Mansurah, Select A State Or Province, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zhu N, Zhang D, Wang W, Li X, Yang B, Song J, Zhao X, Huang B, Shi W, Lu R, Niu P, Zhan F, Ma X, Wang D, Xu W, Wu G, Gao GF, Tan W; China Novel Coronavirus Investigating and Research Team. A Novel Coronavirus from Patients with Pneumonia in China, 2019. N Engl J Med. 2020 Feb 20;382(8):727-733. doi: 10.1056/NEJMoa2001017. Epub 2020 Jan 24. PMID 31978945
- [Result] Cui J, Li F, Shi ZL. Origin and evolution of pathogenic coronaviruses. Nat Rev Microbiol. 2019 Mar;17(3):181-192. doi: 10.1038/s41579-018-0118-9. PMID 30531947
- [Result] Rossignol JF. Nitazoxanide: a first-in-class broad-spectrum antiviral agent. Antiviral Res. 2014 Oct;110:94-103. doi: 10.1016/j.antiviral.2014.07.014. Epub 2014 Aug 7. PMID 25108173
- [Result] Graci JD, Cameron CE. Mechanisms of action of ribavirin against distinct viruses. Rev Med Virol. 2006 Jan-Feb;16(1):37-48. doi: 10.1002/rmv.483. PMID 16287208
- [Result] Caly L, Druce JD, Catton MG, Jans DA, Wagstaff KM. The FDA-approved drug ivermectin inhibits the replication of SARS-CoV-2 in vitro. Antiviral Res. 2020 Jun;178:104787. doi: 10.1016/j.antiviral.2020.104787. Epub 2020 Apr 3. PMID 32251768